CLINICAL TRIAL: NCT04657016
Title: Efficacy and Safety of Tirzepatide Once Weekly Versus Placebo After an Intensive Lifestyle Program in Participants Without Type 2 Diabetes Who Have Obesity or Are Overweight With Weight-Related Comorbidities: A Randomized, Double Blind, Placebo-Controlled Trial (SURMOUNT-3)
Brief Title: A Study of Tirzepatide (LY3298176) In Participants After A Lifestyle Weight Loss Program
Acronym: SURMOUNT-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17246; I8F-MC-GPHM (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-01; First posted 2020-12-07 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Overweight
Keywords: Diet; Exercise; Metabolism and Nutrition Disorder; Behavioral Modification
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Nutrition Disorders | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Participants received weekly doses of tirzepatide subcutaneously (SC) for 72 weeks, starting at 2.5 milligrams (mg) for 4 weeks. Subsequently, the dose was increased by 2.5 mg every 4 weeks up to the maximum tolerated dose (MTD) of either 10 mg or 15 mg.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received matching placebo SC once weekly (QW).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Other: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This is a study of tirzepatide in participants with obesity. The purpose of this study is to learn more about how tirzepatide maintains body weight or adds to weight loss after an intensive lifestyle modification program. The study will last about 2 years (29 visits).

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) ≥30 kg/m2 or ≥27 kg/m2 and previously diagnosed with at least 1 of the following comorbidities: hypertension, dyslipidemia, obstructive sleep apnea or cardiovascular disease
* History of at least one unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Diabetes mellitus
* Change in body weight greater than 5 kg within 3 months prior to starting study
* Obesity induced by other endocrinologic disorders or monogenetic or syndromic forms of obesity
* History of pancreatitis
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Any lifetime history of a suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (65):
- United States (45):
  - National Research Institute - Huntington Park, Huntington Park, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - National Research Institute (NRI) - Santa Ana, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - New Horizon Research Center, Miami, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Elite Clinical Trials, Blackfoot, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Elite Clinical Trials, Rexburg, Idaho
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - American Health Network of IN, LLC, Avon, Indiana
  - American Health Network of IN, LLC, Franklin, Indiana
  - American Health Network of IN, LLC, Muncie, Indiana
  - Cotton O'Neil Mulvane, Topeka, Kansas
  - Tandem Clinical Research,LLC, Marrero, Louisiana
  - The National Diabetes & Obesity Research Institute, Biloxi, Mississippi
  - Clinvest Research LLC, Springfield, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center (WFUBMC), Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Intend Research, LLC, Norman, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Detweiler Family Medicine & Associates, Lansdale, Pennsylvania
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Vanderbilt Health One Hundred Oaks, Nashville, Tennessee
  - Dallas Diabetes Research Center, Dallas, Texas
  - Juno Research, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Argentina (9):
  - Centro Médico Viamonte, CABA, Buenos Aires
  - Investigaciones Medicas Imoba Srl, CABA, Buenos Aires
  - Instituto Centenario, CABA, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Stat Research S.A., Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Glenny Corp, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - CEMEDIAB, C.a.b.a., Ciudad Autónoma de Buenos Aire
  - Instituto Médico Especializado (IME), Buenos Aires
  - Sanatorio Norte, Santiago del Estero
- Brazil (8):
  - CEDOES, Vitória, Espírito Santo
  - Cline Research Center, Curitiba, Paraná
  - Quanta Diagnóstico e Terapia, Curitiba, Paraná
  - CPCLIN, São Paulo, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Puerto Rico (3):
  - Advanced Clinical Research, LLC, Bayamón
  - Manati Center for Clinical Research, Manatí
  - Ponce Medical School Foundation Inc., Ponce

IPD SHARING:
Plan to Share IPD: Yes
Plan Description:
  Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: Access Criteria:
  A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Almandoz JP, Pickett-Blakely O, Tewksbury C, Stefanski A, Gonsahn-Bollie S, Dimitriadis GK, Murro AL, Cao D, Meng Q, Neff LM. Nutritional status with tirzepatide in obesity: A post hoc analysis of the SURMOUNT-1-4 randomized clinical trials. Obes Pillars. 2026 Jan 23;17:100248. doi: 10.1016/j.obpill.2026.100248. eCollection 2026 Mar. PMID 41640675
- [Derived] Wadden TA, Oquendo MA, Kushner RF, Cao D, Karanikas CA, Kechter A, Murphy MA. Psychiatric Safety of Tirzepatide in People With Obesity and No Known Major Psychopathology: A Post Hoc Analysis of SURMOUNT. Obesity (Silver Spring). 2026 Jan 15. doi: 10.1002/oby.70122. Online ahead of print. PMID 41537305
- [Derived] Li X, Cao D, Sapin H, Wang F, Hunter Gibble T, Raibulet NK, Denning M, Kaplan LM. People With Lowest Physical Functioning Scores Showed Greatest Improvement After Tirzepatide Treatment. Obesity (Silver Spring). 2026 Jan;34(1):114-126. doi: 10.1002/oby.70067. Epub 2025 Nov 4. PMID 41187013
- [Derived] Gourgari E, Srivastava G, Kelly AS, Mojdami D, Cao D, Murphy MA, Karanikas CA, Lee CJ. Early-Onset Obesity and Tirzepatide Treatment: A Post Hoc Analysis of the SURMOUNT Clinical Trials. Obesity (Silver Spring). 2025 Sep;33(9):1668-1679. doi: 10.1002/oby.24348. Epub 2025 Jul 27. PMID 40717199
- [Derived] Wadden TA, Chao AM, Machineni S, Kushner R, Ard J, Srivastava G, Halpern B, Zhang S, Chen J, Bunck MC, Ahmad NN, Forrester T. Tirzepatide after intensive lifestyle intervention in adults with overweight or obesity: the SURMOUNT-3 phase 3 trial. Nat Med. 2023 Nov;29(11):2909-2918. doi: 10.1038/s41591-023-02597-w. Epub 2023 Oct 15. PMID 37840095
- See also: A Study of Tirzepatide (LY3298176) In Participants After A Lifestyle Weight Loss Program (SURMOUNT-3) — https://trials.lillytrialguide.com/en-US/trial/1ZuH7WHjpse8JDpVFSSi1I

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a 12-week lead-in period wherein the participants underwent intensive lifestyle modification program to reduce their daily caloric energy intake and increase their physical activity, followed by which they were randomized to receive Tirzepatide or Placebo.
Groups:
- Placebo: Participants received matching placebo subcutaneously (SC) once weekly (QW).
- Tirzepatide: Participants received weekly doses of tirzepatide SC for 72 weeks, starting at 2.5 milligrams (mg) for 4 weeks. Subsequently, the dose was increased by 2.5 mg every 4 weeks up to the maximum tolerated dose (MTD) of either 10 mg or 15 mg.
Period: Overall Study
Arm/Group | Placebo | Tirzepatide
Started | 292 | 287
Received at Least One Dose of Study Drug | 292 | 287
Completed | 227 | 252
Not Completed | 65 | 35
Not completed — Adverse Event | 2 | 4
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 24 | 12
Not completed — Physician Decision | 1 | 2
Not completed — Pregnancy | 2 | 2
Not completed — Protocol Deviation | 1 | 0
Not completed — Withdrawal by Subject | 28 | 14
Not completed — Other - as reported by the investigator | 6 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants received matching placebo SC QW.
- Tirzepatide: Participants received weekly doses of tirzepatide SC for 72 weeks, starting at 2.5 mg for 4 weeks. Subsequently, the dose was increased by 2.5 mg every 4 weeks up to the MTD of either 10 mg or 15 mg.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tirzepatide | Total
Number analyzed (Participants) | 292 | 287 | 579
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.70 (11.79) | 45.40 (12.59) | 45.60 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 181 | 364
  Male | 109 | 106 | 215
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 161 | 151 | 312
  Not Hispanic or Latino | 129 | 132 | 261
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 31 | 63
  White | 252 | 246 | 498
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 44 | 43 | 87
  Brazil | 60 | 59 | 119
  United States | 188 | 185 | 373
Body weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 101.29 (20.67) | 102.47 (22.11) | 101.87 (21.39)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight
Description: Percent change from baseline in body weight. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: All randomly assigned participants who took at least 1 dose of study drug, had a baseline and at least 1 post- baseline value for this outcome, excluding data after discontinuation of study drug.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Placebo: Participants received matching placebo SC once weekly QW.
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
Percent change | 3.3 (0.60) | -21.1 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -24.5, 95% CI 2-sided [-26.1 to -22.8]

2. Primary Outcome: Percentage of Participants With Greater Than or Equal to (≥) 5% Body Weight Reduction
Description: Percentage of participants with ≥5% body weight reduction was analysed by Logistic regression model using imputed data with baseline body weight, Analysis Country, Sex, Treatment as factors.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
percentage of participants | 10.65 | 94.37
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 130.36, 95% CI 2-sided [69.98 to 242.84]

3. Secondary Outcome: Percentage of Participants Who Maintain ≥80% of the Body Weight Lost During Intensive Lifestyle Program
Description: Percentage of participants who maintain ≥80% of the body weight lost during intensive lifestyle program was analysed by logistic regression model using imputed data with baseline body weight, analysis country, sex, treatment as factors.
Time Frame: 72 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
percentage of participants | 37.80 | 98.59
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 101.60, 95% CI 2-sided [39.17 to 263.55]

4. Secondary Outcome: Percentage of Participants Who Achieve ≥10%Body Weight Reduction
Description: Percentage of participants who achieve ≥10% body weight reduction was analysed by logistic regression model using imputed data with baseline body weight, analysis country, sex, treatment as factors.
Time Frame: 72 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
percentage of participants | 4.81 | 88.03
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 153.95, 95% CI 2-sided [78.90 to 300.37]

5. Secondary Outcome: Percentage of Participants Who Achieve ≥15% Body Weight Reduction
Description: Percentage of participants who achieve ≥15% body weight reduction was analysed by logistic regression model using imputed data with baseline body weight, analysis country, sex, treatment as factors.
Time Frame: 72 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
Percentage of participants | 2.06 | 73.94
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 144.48, 95% CI 2-sided [62.65 to 333.21]

6. Secondary Outcome: Percentage of Participants Who Achieve ≥20% Body Weight Reduction
Description: Percentage of participants who achieve ≥20% body weight reduction was analysed by logistic regression model using imputed data with baseline body weight, analysis country, sex, treatment as factors.
Time Frame: 72 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
Percentage of participants | 1.03 | 54.93
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 118.06, 95% CI 2-sided [40.08 to 347.74]

7. Secondary Outcome: Change From Baseline in Waist Circumference
Description: Change from baseline in waist circumference. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Centimeters (Cms)
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
Centimeters (Cms) | 1.1 (0.58) | -16.8 (0.56)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -17.9, 95% CI 2-sided [-19.5 to -16.3]

8. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
kg | 3.5 (0.67) | -21.5 (0.65)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -25.0, 95% CI 2-sided [-26.9 to -23.2]

9. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change from baseline in BMI. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilogram per meter square (kg/m^2)
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
kilogram per meter square (kg/m^2) | 1.2 (0.23) | -7.7 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -8.9, 95% CI 2-sided [-9.6 to -8.3]

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Description: Change from baseline in SBP. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
millimeters of mercury (mmHg) | 4.4 (0.76) | -5.8 (0.73)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -10.2, 95% CI 2-sided [-12.2 to -8.1]

11. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP)
Description: Change from baseline in DBP. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 291 | 284
mmHg | 2.3 (0.53) | -3.4 (0.51)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -5.7, 95% CI 2-sided [-7.2 to -4.3]

12. Secondary Outcome: Percent Change From Baseline in Total Cholesterol
Description: Percent change from baseline in total cholesterol. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 252 | 263
Percent change | 5.19 (1.11) | -3.00 (0.97)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -7.79, 95% CI 2-sided [-10.40 to -5.10], Standard Error of Mean 1.348

13. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein (HDL) Cholesterol
Description: Percent change from baseline in HDL cholesterol. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 252 | 263
Percent change | 3.6 (1.12) | 15.4 (1.19)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 11.4, 95% CI 2-sided [8.2 to 14.7], Standard Error of Mean 1.67

14. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein (LDL) Cholesterol
Description: Percent change from baseline in LDL cholesterol. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 252 | 263
Percent change | 6.14 (1.71) | -6.07 (1.44)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -11.50, 95% CI 2-sided [-15.30 to -7.53], Standard Error of Mean 1.97

15. Secondary Outcome: Percent Change From Baseline in Very Low-Density Lipoprotein (VLDL) Cholesterol
Description: Percent change from baseline in VLDL cholesterol. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 252 | 261
Percent change | 3.0 (2.32) | -25.6 (1.60)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -27.8, 95% CI 2-sided [-32.1 to -23.2], Standard Error of Mean 2.25

16. Secondary Outcome: Percent Change From Baseline in Triglycerides
Description: Percent change from baseline in triglycerides. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 252 | 263
Percent change | 3.0 (2.34) | -25.8 (1.61)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -28.0, 95% CI 2-sided [-32.3 to -23.4], Standard Error of Mean 2.26

17. Secondary Outcome: Percent Change From Baseline in Free Fatty Acids
Description: Percent change from baseline in free fatty acids. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 251 | 263
Percent change | -15.0 (2.95) | -33.1 (2.20)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -21.3, 95% CI 2-sided [-28.4 to -13.6], Standard Error of Mean 3.76

18. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Change from baseline in fasting glucose. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Milligram per deciliter (mg/dL)
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 276 | 275
Milligram per deciliter (mg/dL) | 2.4 (0.86) | -8.8 (0.82)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -11.2, 95% CI 2-sided [-13.5 to -8.8]

19. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 275 | 278
Percentage of HbA1c | 0.01 (0.022) | -0.46 (0.020)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.47, 95% CI 2-sided [-0.53 to -0.42]

20. Secondary Outcome: Percent Change From Baseline in Fasting Insulin
Description: Percent change from baseline in fasting insulin. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Analysis Country + Sex + Lead-In Weight Loss % + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 275 | 277
Percent change | 17.3 (4.95) | -39.1 (2.46)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -48.1, 95% CI 2-sided [-53.7 to -41.7], Standard Error of Mean 3.04

21. Secondary Outcome: Change From Baseline in Short Form 36 Version 2 Health Survey Version 2 (SF 36v2) Acute Form Physical Functioning Domain Score
Description: The SF-36v2 acute form assesses health-related quality of life (HRQoL) on 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The Physical-Functioning domain assesses limitations due to health "now" and consists of 10-items, each rated on a 3-point Likert scale. Scoring of the domain is norm-based and presented in the form of T-scores, with a mean of 50 and standard deviation of 10; higher scores indicate better levels of function. Range cannot be specified in norm-based scores.
  LS mean was determined using analysis of covariance (ANCOVA) model using Baseline + Analysis Country + Sex + Lead-In Weight Loss % + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 209 | 231
T-score | -0.6 (0.39) | 3.3 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 3.8, 95% CI 2-sided [2.8 to 4.9]

22. Secondary Outcome: Change From Baseline in Impact of Weight on Quality of Life Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score
Description: The IWQOL Lite-CT consists of 20 items, assessing 2 primary domains of obesity related HRQoL: Physical (7 items) and Psychosocial (13 items). A 5-item subset of the Physical domain - the Physical Function composite - is also supported. Items in the Physical Function composite describe physical impacts related to general and specific physical activities. All items in the physical domain are rated on either a 5-point frequency ("never" to "always") scale or a 5-point truth ("not at all true" to "completely true") scale. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better health-related quality of life.
  LS mean was determined using ANCOVA model with Baseline + Analysis Country + Sex + Lead-In Weight Loss % + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, 72 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 201 | 226
score on a scale | 1.1 (1.17) | 13.9 (1.10)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 12.8, 95% CI 2-sided [9.7 to 16.0]

ADVERSE EVENTS:
Time Frame: Baseline up to week 76
Description: All randomized participants who received at least one dose of study drug. Based on the planned safety analysis, adverse events were collected per the treatment regimen, irrespective of each dose level.
Arm/Group | Placebo | Tirzepatide
All-Cause Mortality (participants affected / at risk) | 1/292 | 1/287
Serious Adverse Events (participants affected / at risk) | 14/292 | 17/287
Other Adverse Events (participants affected / at risk) | 172/292 | 230/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=292) | Tirzepatide (N=287)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (3) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=292) | Tirzepatide (N=287)
Abdominal pain (Gastrointestinal disorders) | 7 (10) | 30 (38)
Constipation (Gastrointestinal disorders) | 20 (24) | 66 (89)
Diarrhoea (Gastrointestinal disorders) | 27 (53) | 89 (233)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 27 (47)
Eructation (Gastrointestinal disorders) | 3 (3) | 16 (26)
Flatulence (Gastrointestinal disorders) | 8 (8) | 19 (24)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (9) | 19 (44)
Nausea (Gastrointestinal disorders) | 41 (112) | 114 (499)
Vomiting (Gastrointestinal disorders) | 4 (4) | 52 (133)
Fatigue (General disorders) | 9 (9) | 20 (23)
Injection site reaction (General disorders) | 3 (3) | 32 (204)
Covid-19 (Infections and infestations) | 74 (80) | 66 (69)
Influenza (Infections and infestations) | 25 (30) | 12 (13)
Sinusitis (Infections and infestations) | 16 (18) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 21 (32) | 25 (37)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13) | 27 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (16) | 17 (19)
Dizziness (Nervous system disorders) | 6 (6) | 20 (24)
Headache (Nervous system disorders) | 22 (27) | 27 (37)
Anxiety (Psychiatric disorders) | 19 (19) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT04657016/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT04657016/SAP_001.pdf